CLINICAL TRIAL: NCT05263674
Title: Fast Acute Sedation at Intensive Care vs. High-dose i.v. Anti-seizure Medication for Treatment of Non-convulsive Status Epilepticus (FAST-trial)
Acronym: FAST
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Aarhus University Hospital (Other); University Hospital of Zealand (Unknown); Copenhagen University Hospital, Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21/34684; 2021-003392-34 (EudraCT Number)
Record Dates: First submitted 2022-01-17; First posted 2022-03-02 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Non-Convulsive Status Epilepticus
MeSH Terms: conditions — Status Epilepticus

STUDY DESIGN:
Intervention Model Description: Comparison of two treatment strategies
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- "Non-sedative medical treatment" (No Intervention): The patient is treated with an additional high-dose intravenous antiepileptic drug, which is selected by the treating neurologist. If NCSE continues to be detected at cEEG or clinically> 3 hours after starting treatment, the patient should receive standard treatment (i.e. sedation in the intensive care unit or addition of additional intravenous antiepileptic drugs) in accordance with local guidelines and the assessment of the treating neurologist. The following preparations are permitted as additional treatment:
  Levetiracetam (60 mg / kg as saturation dose followed by maintenance dose of 2-4 g / day), valproate (60 mg / kg as saturation dose followed by maintenance dose of 20 mg / kg / day), phosphenytoin (20 PE as saturation dose followed by maintenance dose 5 mg PE / kg / day), lacosamide (400 mg as a saturation dose followed by a maintenance dose of 200-400 mg / day), topiramate (200-400 mg per probe as a saturation dose followed by a maintenance dose of 200-400 mg / day).
- Fast sedation (Experimental): Within a maximum of 60 minutes after the diagnosis of NCSE (EEG or clinical), the patient must be sedated with high-dose Propofol (bolus 3-5 g / kg, maintenance dose 5-10 mg / kg / hour) to - 5 on the Richmond agitation sedation scale (RASS) for 20 hours, and a single anti-epileptic drug should be added as adjunctive therapy. Addition of low-dose Midazolam (max. 0.1 mg / kg / h) is permitted if deep sedation (defined clinically by RASS -5) is not possible with Propofol alone. After 20 hours, the sedation should be completely phased out within 3 hours.
  Interventions: Drug: Rapid sedation

INTERVENTIONS:
Drug: Rapid sedation — High-dose Propofol (bolus 3-5 g / kg, maintenance dose 5-10 mg / kg / hour) to - 5 on the Richmond agitation sedation scale (RASS) for 20 hours, and a single anti-epileptic drug should be added as adjunctive therapy. Addition of low-dose Midazolam (max. 0.1 mg / kg / h) is permitted if deep sedation (defined clinically by RASS -5) is not possible with Propofol alone.
  Arms: Fast sedation

SUMMARY:
This open-label, randomized multicenter trial aims at clarifying the standard of care of patients with non-convulsive status epilepticus not responding to treatment with benzodiazepines and at least one high-dose intra venous anti-seizure medication.

DETAILED DESCRIPTION:
Persistent epileptic seizures, aka. status epilepticus (SE), are the second most common neurological cause of acute admissions. Around halv of the patients suffers from SE without prominent visible seizures ("convulsions"), which is referred to as non-convulsive status epilepticus (NCSE) and is afflicted with a long-term mortality of >50% also in patients without concomittant acute brain disease. There are no evidence-based treatment guidelines for NCSE but patients usually receive treatment with benzodiazepines followed by i.v. anti-seizure medication. If seizures continues, further treatment is controversial. The participating centers have long-standing experience in treating NCSE but use different, internationally accepted treatment strategies. Some initiate aggressive treatment with fast sedation at intensive care aiming at immediate seizure control, other estimate that the side effects of sediation does not outweigh the potential benefit and try high-dose i.v. anti-seizure medication that only slightly impair conciousness - often with success.

This randomized, open label, multicenter trial (Eudract 2021-003392-34) aims at clarifying the treatment of patients with NSCE not responding to standard therapy. Patients with verified NCSE based on clinical parameter or using electroencephalography (EEG) are randomized into a fast acute sedation group and a group that receives at least one additional, high-dose anti-seizure mediciation.

Primary objective endpoint is treatment failure 24 h after randomization as determined by EEG. Secondary endpoints are e.g. seizure-induced neurological damage, treatment-related complications and neurological long-term outcome.

The statistical planing aims at showing superiority of aggressive treatment, 140 patients shall be included in a three years period at the University Hospitals in Aarhus, Odense, Roskilde and Copenhagen.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (older than 18 years) with EEG-verified NCSE, according to the Salzburg criteria, who have not responded to appropriate treatment with benzodiazepines and at least one 2nd line i.v. anti-seizure medication according to the current Danish national neurological treatment guidelines (Levetiracetam, Fosfenytoin or Valproate).

Exclusion Criteria:

* patients with epilepticus status due to acute neuroinfection (e.g. bacterial meningitis or viral encephalitis)
* acute traumatic or spontaneous intracranial hemorrhage
* suspicion of cerebral anoxia / hypoxia / hypoglycemia / epileptic encephalopathy
* contraindications to anti-seizure medication defined in the protocol
* contraindications to anesthesia treatment in intensive care
* focal motor status epilepticus without relevant conscious influence (Glasgow Coma Scale> 13)
* known epileptic encephalopathy
* Clinical need for acute intubation

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-02-07 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with continued NCSE on EEG after 24 h ("treatment failure") | 24 hours after randomisation
  NCSE diagnosed using EEG and defined by the "Salzburg criteria" for NCSE (e.g. Leitinger et al. Lancet Neurology, 2016)

SECONDARY OUTCOMES:
Number of treatment related complications | at discharge, on average after 7 days
  e.g. tracheostoma, infections
New neurological deficit | at discharge, on average after 7 days
  Neurological deficits are quantified using National Institute of Health Stroke Scale (NIHSS, maximum possible score is 42, the minimum score - indicating no deficits - is 0) at admission and discharge. New neurological deficit is defined as increase of NIHSS >5 at discharge

OTHER OUTCOMES:
Influence of cEEG on new neurological deficit | at discharge, on average after 7 days
  Patients receive either cEEG or spot EEG depending on the center. In this pre-specified analyses, the impact of cEEG vs. spot-EEG on the degree of new neurological deficits (outcome 3) will be compared
Duration of intensive care treatment | at discharge, on average after 7 days
  Definition: Time from intubation to discharge from ICU
Duration of hospitalization | 1-100 days, on average 7 days
  Time from randomization to discharge from hospital in charge for acute treatment of NCSE
Proportion of patients with superrefractory status epilepticus | at discharge, on average after 7 days
  Proportion of patients that develop superrefractory status epilepticus after randomization but during current hospitalization
Survival after discharge | 3, 6, 12, and 24 months after randomization
  Determined at ambulatory control 3,6,12 and 24 months after randomization
Quality of life after discharge | 3, 6, 12, and 24 months after randomization
  Determined using questionnaire/patient survey (Quality of Life in Epilepsy Inventory, Qolie-31 Danish translation), at ambulatory controls 3, 6, 12, and 24 months after randomization

CONTACTS AND LOCATIONS:
Locations (4):
- Denmark (4):
  - Aarhus Universitetshospital, Aarhus
  - Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense
  - University Hospital of Zealand, Roskilde

IPD SHARING:
Plan to Share IPD: No
Anonymized IPD will be shared upon reasonable request within the limits of Danish legislation for data security.

REFERENCES:
- [Derived] Cornwall CD, Piilgaard H, Engedal TS, Olsen HT, Moller K, Kroigard T, Uslu B, Christensen J, Sidaros A, Beier CP. Fast Acute Sedation at Intensive Care vs. High-Dose IV Anti-seizure Medication for Treatment of Non-convulsive Status Epilepticus: A Randomized, Multicenter Trial. Crit Care Explor. 2025 Sep 15;7(9):e1311. doi: 10.1097/CCE.0000000000001311. eCollection 2025 Sep 1. PMID 40953286